CLINICAL TRIAL: NCT06879223
Title: Effect of Oral Health Educational Program on the Oral Health-Related Quality of Life in a Group of Children with Chronic Kidney Disease: a Before and After Pilot Study
Brief Title: Effect of Oral Health Educational Program on the Oral Health Related Quality of Life in a Group of Children with Chronic Kidney Disease
Acronym: CKD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hebaallah Samy Gamil Mohamed, Dentist, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Educational program on CKD
Record Dates: First submitted 2025-03-10; First posted 2025-03-17 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Chronic Kidney Disease(CKD)
Keywords: CKD OHRQL; OHEP
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Children with CKD (Experimental)
  Interventions: Behavioral: Oral Health Educational Program

INTERVENTIONS:
Behavioral: Oral Health Educational Program — Providing the children with an educational program through a data show presentation when and how to brush their teeth, causes of dental caries and how to prevent its occurrence. A flyer will be distributed including simple language about preventive measure of dental caries and schedule of teeth brushing to ensure retention of information.

SUMMARY:
Children with CKD are at higher risk for poor oral health28 due to factors such as compromised immunity, medication side effects, and dietary restrictions. Poor oral health can lead to pain, infection, and difficulties in eating and speaking, which in turn negatively affects their quality of life. This study is designed to address this gap by exploring how an oral health educational program could improve the oral health-related quality of life (OHRQoL) in this group.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-10 years old.
* Diagnosed with Chronic Kidney Disease

Exclusion Criteria:

* Children with other systemic diseases.
* Parents that refuse the participation of their children.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-06-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Oral health related quality of life | 3 months
  it will be assessed using a questionnaire and the measurement unit is percentage

SECONDARY OUTCOMES:
Developmental enamel defect. | 3 months
  it will be assessed using the DDE (Developmental Defects of Enamel) index and the measurement unit is Mean SD.
  The DDE index categorizes defects into three main types:
  Opacities: Changes in enamel translucency, which can be diffuse or demarcated. Hypoplasia: A quantitative defect where enamel is thinner or missing in certain areas.
  Discoloration: Changes in enamel color due to structural abnormalities. higher scores means worse outcome.
Caries experience. | 3 months
  it will be assessed using the def(decayed, extracted,filled) index and the measurement unit is Mean SD.
  The def score is the sum of these values, providing an indication of oral health in children before their permanent teeth emerge.
  higher scores means worse outcome.
Caries experience | 3 months
  it will be assessed using the DMF (Decayed, Missing, Filled) index and the measurement unit is mean SD.
  The DMF score is the sum of these values, indicating the overall caries experience in an individual or population. Unlike the def index, which applies to primary teeth, the DMF index is used for permanent teeth.
  higher scores means worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo Unversity, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Undecided